CLINICAL TRIAL: NCT04340908
Title: Effects of SGLT2 Inhibitor on Type 2 Diabetic Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongchang Guo (Other)
Responsible Party: Sponsor-Investigator, Hongchang Guo, Attending doctor, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ-SGLT2i
Record Dates: First submitted 2020-04-02; First posted 2020-04-10 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2; Cardiac Surgery
Keywords: Diabetes Mellitus; Outcome; SGLT2 inhibitors; Cardiac Surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Dapagliflozin 10 mg tablet
  Interventions: Drug: Dapagliflozin 10 MG
- Control (Placebo Comparator): matching placebo tablet
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — 10 mg tablet, oral, once daily, 1-year treatment, postoperation
  Other Names: Forxiga
  Arms: Treatment
Drug: Placebos — matching placebo tablet, oral, once daily, 1-year treatment, postoperation
  Arms: Control

SUMMARY:
Patients with diabetes have poorer cardiac surgery outcomes compared with non-diabetics. Proper blood glucose management is critical to reduce the morbidity and mortality for diabetic patients after cardiac surgery.

SGLT2 inhibitors including dapagliflozin as a new diabetes drug can reduce heart failure hospitalization rates and overall cardiovascular mortality in patients with cardiovascular disease.

This study is to assess the impact of one year of treatment of SGLT2 inhibitors on cardiac function, postoperative complications and long-term cardiovascular mortality in diabetic patients undergoing cardiac surgery.

The investigators use echocardiography to evaluated cardiac function in diabetic patients during perioperative cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at index date.
2. Diagnosis of Type 2 Diabetes.
3. Scheduled for cardiac surgery (coronary artery bypass grafting, valve replacement, ventricular assist device, cardiac transplantation, or any other surgery requiring thoracotomy).
4. eGFR ≥ 60 ml/min/1.73 m2.
5. Patients who agree to receive treatment with SGLT2 inhibitors.
6. Patients must be on current stable hemodynamic profile , without dehydration.

Exclusion Criteria:

1. Diagnosis of Type 1 Diabetes.
2. eGFR < 60 ml/min/1.73 m2.
3. Unstable or rapidly progressive renal disease.
4. Hypersensitivity to dapagliflozin or any excipients.
5. Severe hepatic disease.
6. Patients who have participated in any other clinical trial of an investigational medicinal product within the previous 30 days.
7. Any other reason considered by a study physician to be inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in mean EF% between the treatment and control study arms | 2 year
  Echocardiography is used to assess cardiac function.
Difference in NTproBNP between the treatment and control study arms | 2 year
  NT-proBNP is used to assess cardiac function.

SECONDARY OUTCOMES:
All-cause postoperative mortality | 2 year
  All-cause mortality identified during two years follow-up.
Rehospitalization for cardiovascular causes | 2 year
  Rehospitalization due to cardiovascular diseases during two years follow-up.
Serious postoperative infection | 2 year
  Including postoperative sternal dehiscence, external genital infections, etc.
Acute postoperative kidney injury | 2 year
  Acute postoperative kidney injury requiring renal replacement therapy
Hypoglycemia | 2 year
  Identified using ICD9 and ICD10 codes and reported as rates.
Duration of Hospitalization | 2 year
  Days from date of surgery to hospital discharge.
Diabetic ketoacidosis | 2 year
  Identified using ICD9 and ICD10 codes and reported as rates.
Lactic acidosis | 2 year
  Identified using ICD9 and ICD10 codes and reported as rates.
Post operative atrial fibrillation | 7 days
  In this study, postoperative AF was defined as occurrence of the arrhythmia within the first 7 days after cardiac surgery. AF was considered to be present when an irregular rhythm was detected in the absence of P waves and/or an f wave was detected.

CONTACTS AND LOCATIONS:
Overall Officials: Lai, M.D., Study Chair — Beijing Anzhen Hospital; Guo, M.D., Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Mediacal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No